CLINICAL TRIAL: NCT04443595
Title: Dual-scopic Pancreatic Necrosectomy (DPN): Laparoscopic Pancreatic Necrosectomy (LPN) and Nephroscopic Pancreatic Necrosectomy (NPN)
Brief Title: Dual-scopic Pancreatic Necrosectomy (DPN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Yang Cai, Director, Deputy Chief of Hepatobiliary and Pancreatic Surgery, Professor., First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-009-1
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Pancreatitis; Pancreatitis, Acute Necrotizing; Pancreatic Diseases
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Acute Necrotizing; Pancreatic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Treatment of Acute Severe Pancreatitis with DPN
  Interventions: Procedure: Dual-scopic pancreatic necrosectomy（DPN）

INTERVENTIONS:
Procedure: Dual-scopic pancreatic necrosectomy（DPN） — Treatment of Acute Severe Pancreatitis with DPN

SUMMARY:
The LPN procedure is performed under general anesthesia. The transperitoneal access to peripancreatic space is via the gastro-colic ligament and greater omentum, effusion and pus is removed by laparoscopic forceps and suction. Laparoscopic cholecystectomy (LC) is performed during the LPN procedure on patients with indication.

The NPN procedure is followed by the standard retroperitoneal approach. After the catheter is exchanged over a guide wire and serially dilated up from 6F to 24F followed by Seldinger technique, the access track to the necrotic cavity is established. A nephroscope is inserted into the cavity through the track for debridement. Using forceps and suction, the peripancreatic solid necrotic tissue and pus is grasped and removed. A large-bore irrigating drain is left in the cavity, with continuous irrigation by warm normal saline solution at a rate of 100-125 ml/h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 18 or above admitted to UPMC with a diagnosis of AP based on at least 2 of the following criteria:(i) abdominal pain characteristic of AP (ii) serum amylase and/or lipase ≥ 3 times the upper limit of normal (iii) characteristic findings of AP on abdominal CT scan will be screened for study enrollment.

Exclusion Criteria:

* Less than 18 years of age
* Pregnant women
* Presence of renal dysfunction (Cr>1.5mg/dL)
* Pre existing heart dysfunction or NYHA classification score above III
* Coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication Rate | through study completion, an average of 24 weeks
  Proportion of patients with perioperative complications
Mortality | through study completion, an average of 24 weeks
  Proportion of patients dying in the perioperative period

SECONDARY OUTCOMES:
Hospital stay | through study completion, an average of 24 weeks
  Length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No